CLINICAL TRIAL: NCT02547948
Title: CD19-targeting CAR T Cells for Refractory B Cell Lymphoma
Brief Title: CD19-targeting CAR T Cells for B Cell Lymphoma
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fuda Cancer Hospital, Guangzhou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CD19-targeting CAR T
Record Dates: First submitted 2015-09-04; First posted 2015-09-14 (Estimated); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: B Cell Lymphoma
Keywords: CD19; CAR T Cells; Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CAR T cells (Experimental): In interventional studies, participants are assigned to accept CD19-targeting CAR T Cells infusion so that researchers can evaluate the effects of the interventions on biomedical or health-related outcomes. Arm refers to each group or subgroup of participants in a clinical trial that receives specfic interventions (or no intervention) according to the study protocol. This is decided before the trial begins.
  Interventions: Biological: CD19-targeting CAR T Cells infusion
- No Intervention (No Intervention)

INTERVENTIONS:
Biological: CD19-targeting CAR T Cells infusion — CD19-targeting 2nd generation CAR t cells infusion for refractory B cell lymphoma
  Arms: CAR T cells

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of CD19-targeting CAR T Cells infusion for B Cell Lymphoma.

DETAILED DESCRIPTION:
Chimeric antigen receptor (CAR) T cells targeting CD19 will be evaluated for safety and efficacy in patients with B cell lymphoma or leukemia. The CAR consists of a CD19 targeting antibody scFv with two intracellular signaling domains derived from CD3 zeta and CD28. Autologous T cells will be gene-engineered with the CAR gene using a retrovirus vector. Prior to T cell infusion, the patients will be subjected to preconditioning treatment. After T cell infusion, the patients will be evaluated for 24 months for adverse reactions, persistence of CAR T cells and efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Relapsed or refractory CD19+ B-cell lymphoma.
2. Measurable disease.
3. Performance status ECOG 0-2.
4. Age:18-80.
5. Fertile females/males must consent to use contraceptives during participation of the trial.
6. Signed informed consent

Exclusion Criteria:

1. Any significant medical or psychiatric illness that would prevent the patient from giving informed consent or from following the study procedures.
2. Patients with primary CNS lymphoma.
3. Known human immunodeficiency virus (HIV) infection.
4. Active and/or severe infection (e.g. tuberculosis, sepsis and opportunistic infections, active hepatitis B virus (HBV) or active hepatitis C virus (HCV) infection).
5. Other serious underlying medical conditions, which, in the Investigator's judgment, could impair the ability of the patient.
6. Treatment with an investigational product within 30 days prior to enrollment, or at least 5 half lives of that drug, which is longest.
7. Patients that do not consent to that tissue and blood samples are stored in a biobank.
8. Pregnancy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-08-15 (Actual); Study Completion 2016-08-15 (Actual)

PRIMARY OUTCOMES:
CAR T cell persistence | up to 24 months
  Presence of circulating CAR T cells will be evaluated with flow cytometry and real time PCR in patient blood

SECONDARY OUTCOMES:
Tumor load | up to 24 months
  Tumor load will be quantified with radiology, bone marrow and/or blood samples dependent on diagnosis

OTHER OUTCOMES:
B cell number and immunoglobulins | up to 24 months
  Number of blood B cells and immunoglobulins will be evaluated by routine diagnostics

CONTACTS AND LOCATIONS:
Overall Officials: Lizhi Niu, PhD, Study Chair — Fuda Cancer Hospital
Locations (1):
- Central laboratory in Fuda cancer hospital, Guangzhou, Guangdong, China